CLINICAL TRIAL: NCT01419548
Title: An Early Phase 1 Study of ABT-888 in Combination With Carboplatin and Paclitaxel in Patients With Hepatic or Renal Dysfunction and Solid Tumors
Brief Title: ABT-888, Carboplatin, and Paclitaxel for Cancer With Liver or Kidney Problems
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110215; 11-C-0215
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-11-18

CONDITIONS: Neoplasms
Keywords: ABT-888; Liver Dysfunction; Kidney Dysfunction; PARP Inhibitor; Pharmacokinetics; Cancer
MeSH Terms: conditions — Neoplasms; Liver Diseases | interventions — veliparib; Carboplatin; Paclitaxel

INTERVENTIONS:
Drug: ABT-888
Drug: Carboplatin
Drug: Paclitaxel

SUMMARY:
Background:

- Paclitaxel and carboplatin are two standard drugs that stop cancer cells from reproducing. ABT-888 is an experimental cancer drug that may prevent cancer cells from "fixing" the damage done by chemotherapy drugs. This may make the chemotherapy work better. More tests are needed to determine the safety and effectiveness of ABT-888 plus chemotherapy. Researchers also want to find the best dose of ABT-888 for people who have kidney or liver problems in addition to cancer.

Objectives:

- To test the safety and effectiveness of ABT-888 plus carboplatin and paclitaxel in people who have both cancer and kidney or liver problems.

Eligibility:

* Individuals at least 18 years of age who have solid tumors that have not responded to standard treatment, and who also have kidney or liver problems.
* A small group of people with solid tumors and normal kidney and liver function may also receive treatment for study comparison purposes.

Design:

* Participants will be screened with a medical history and physical exam. They will have blood and urine tests, tumor samples, tests of liver and kidney function, and imaging studies. Participants will also provide a hair sample at the start of the study.
* Participants will take one dose of ABT-888 1 week before starting chemotherapy. The two chemotherapy drugs will be given on day 3 of a 21-day cycle. Participants will take ABT-888 daily for the first 7 days of each cycle.
* They will keep a diary to record medication doses and any side effects. They will also have frequent blood tests and imaging studies. Participants will provide more hair samples on day 3 of cycle 1 before and after having paclitaxel.
* Participants will continue treatment for up to 18 weeks as long as the cancer stops growing or shrinks and there are no serious side effects. Participants may have the option to continue treatment after the study is done.

DETAILED DESCRIPTION:
Background:

The poly (ADP-ribose) polymerase (PARP) family of enzymes is critical for maintaining genomic stability by regulating a variety of DNA repair mechanisms. The carboplatin/paclitaxel combination has demonstrated a wide spectrum of clinical antitumor activity, making it an ideal platform for evaluation with novel agents, such as the PARP inhibitor ABT-888.

Objectives:

To determine the pharmacokinetics and pharmacodynamics of ABT-888 in patients with varying degrees of renal or hepatic dysfunction.

To determine the maximum tolerated dose (MTD) of ABT-888 in combination with carboplatin and paclitaxel for patients with varying degrees of liver or kidney dysfunction.

To provide dosing recommendations for ABT-888 in combination with carboplatin and paclitaxel based on degree of hepatic and renal impairment.

To define the dose-limiting toxicity and other toxicities associated with the use of this combination in patients with varying degrees of renal or hepatic dysfunction.

To evaluate the pharmacokinetic parameters of ABT-888, carboplatin and paclitaxel when administered as a combination in patients with varying degrees of renal or hepatic dysfunction.

To evaluate the pharmacodynamic measurement of PAR and platinum adducts in peripheral blood mononuclear cells (PBMC) and tumor cells associated with the use of this combination

in patients with varying degrees of renal or hepatic dysfunction.

Eligibility:

Patients must have histologically confirmed malignancy that is metastatic or unresectable, for which standard curative or palliative measures do not exist or are no longer effective, and for which there is expectation of response to the combination of carboplatin/paclitaxel (e.g., lung, ovarian, breast, and melanoma).

Patients must have adequate bone marrow function.

Patients with normal organ function, patients with all degrees of renal dysfunction, and patients with mild to severe hepatic dysfunction are allowed.

Study Design:

ABT-888 (80 mg) will be given orally on day -6 ( 1 day) of cycle 1 in all cohorts. ABT-888 in varying doses will then be given on days 1-7 of each cycle, with the dose depending on each patient's degree of renal or hepatic dysfunction.

Fixed doses of chemotherapy will be given intravenously on day 3 of each cycle. For patients with renal dysfunction, carboplatin will be given at AUC of 6 and paclitaxel at 175 mg/m2. For patients with hepatic dysfunction, carboplatin will be given at AUC of 6 and paclitaxel at doses adjusted to each patient's degree of hepatic dysfunction.

The dose of ABT-888 will be escalated to determine the MTD of the combination.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed malignancy that is metastatic or unresectable, for which standard curative or palliative measures do not exist or are no longer effective, and for which there is expectation of response to the combination of carboplatin/paclitaxel (e.g., lung, ovarian, breast, melanoma).
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of ABT-888 in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric phase 1 combination trials.
* ECOG performance status less than or equal to 2.
* Life expectancy of greater than 12 weeks.
* Patients must have marrow function as defined below:

absolute neutrophil count greater than or equal to 1,500/mcL

platelets greater than or eqaul to 100,000/mcL

hemoglobin greater than or eqaul to 8.0 g/dL

* Patients with all degrees of renal dysfunction are allowed including patients on hemodialysis. Patients with mild to severe hepatic dysfunction are allowed as defined below:
* total bilirubin less than or eqaul to 5 times ULN AND AST and ALT less than or eqaul to10 times ULN

For patients with a recently placed biliary stent, patients should have consistent results within a hepatic group from two laboratory readings within 3 days apart, taken at least 10 days following biliary stent placement. For patients with a biliary stent placed over 2 months ago, no obstruction or blockage can have occurred within the last 2 months.

-The effects of ABT-888 on the developing human fetus are unknown. For this reason and because other therapeutic agents or modalities used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study

participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

-Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those whose adverse event due to agents administered more than 4 weeks earlier have not resolved or stabilized. Patients who have been administered ABT-888 as part of a single or combination, Phase 0 or I study, should not necessarily be excluded from participating in this study solely because of receiving prior ABT-888.
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888 or other agents used in study.
* Peripheral neuropathy of severity greater than grade 1.
* Inability to take oral medications on a continuous basis.
* Evidence of bleeding diathesis.
* Patients with brain metastasis should have stable disease for at least 4 weeks following therapy for brain metastasis (such as surgery, radiotherapy or stereotactic radiosurgery).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ABT-888 is PARP inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ABT-888, breastfeeding should be discontinued if the mother is treated with ABT-888. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions with ABT-888 as well as possible interactions with paclitaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. However, HIV-positive patients without an AIDS-defining diagnosis who are not receiving agents with the potential for PK interactions with ABT-888 may be eligible.
* Patients with both hepatic and renal dysfunction will also be excluded.
* Patients who received and progressed on the combination of carboplatin/paclitaxel will not be eligible.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-29; Primary Completion 2011-11-18 (Actual); Study Completion 2011-11-18 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetics and pharmacodynamics of ABT-888 in patients with varying degrees of renal or hepatic dysfunction. To determine the MTD of ABT-888 with carboplatin and paclitaxel in these patients.
To determine the pharmacokinetics and pharmacodynamics of ABT-888 in patients with varying degrees of renal or hepatic dysfunction.
To determine the MTD of ABT-888 with carboplatin and paclitaxel in these patients.

SECONDARY OUTCOMES:
To define the dose-limiting toxicity and other toxicities associated with the use of this combination in patients with varying degrees of renal or hepatic dysfunction.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Pittsburgh Cancer Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Ame JC, Spenlehauer C, de Murcia G. The PARP superfamily. Bioessays. 2004 Aug;26(8):882-93. doi: 10.1002/bies.20085. PMID 15273990
- [Background] Shiobara M, Miyazaki M, Ito H, Togawa A, Nakajima N, Nomura F, Morinaga N, Noda M. Enhanced polyadenosine diphosphate-ribosylation in cirrhotic liver and carcinoma tissues in patients with hepatocellular carcinoma. J Gastroenterol Hepatol. 2001 Mar;16(3):338-44. doi: 10.1046/j.1440-1746.2001.02378.x. PMID 11339428
- [Background] Tomoda T, Kurashige T, Moriki T, Yamamoto H, Fujimoto S, Taniguchi T. Enhanced expression of poly(ADP-ribose) synthetase gene in malignant lymphoma. Am J Hematol. 1991 Aug;37(4):223-7. doi: 10.1002/ajh.2830370402. PMID 1907096